CLINICAL TRIAL: NCT05873478
Title: Effects Of High Intensity Interval Training on Cognitve Flexibility Among Female Teenagers
Brief Title: Effects of High Intensity Interval Training on Cognitive Flexibility Among Female Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Professor, Riphah International University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01497
Record Dates: First submitted 2023-02-09; First posted 2023-05-24 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Flexibility Among Female Teenagers
Keywords: Cognitive Flexibility; High Intensity Interval Training; High Intensity Exercises; Digital Span Test; Mini Mental State Examination
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: one group is taking intervention and other is control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (High Intensity Interval Training) (Experimental): High Intensity Interval Training for 8 weeks, which include lunges, squatting sprinting and other exercises.
  Interventions: Other: High Intensity Interval Training
- Control (No Intervention) (No Intervention): Control Group received no intervention they all will be engaged in normal daily routines.

INTERVENTIONS:
Other: High Intensity Interval Training — The HIIT sessions ranging from 4-12 minutes in duration for 8 weeks in which three sessions will be conducted each week (weeks 1-3: 4 minutes; weeks 4-6: 8 minutes; weeks 7-8: 12 minutes respectively), with a work to rest ratio of 30sec: 10sec, as mention in table 1. Experimental group/HIT group engaged in their HIIT sessions (inclusive of a short warm-up activity including dynamic exercises i.e., walking/running, 8-10 minutes of HIIT and cool down which include static exercises i.e., shoulder and hip muscle stretches). Session duration and intensity are increased with weekly progression in intervention groups. The high resistance training sessions was be delivered by the researcher to HIT group
  Arms: Experimental (High Intensity Interval Training)

SUMMARY:
The study suggests that the high intensity exercise training program is beneficial for the female teenagers to enhance their cognitive abilities along with the physical strengthening. It also helps the teenagers to increase their mental health for better health and memory.

DETAILED DESCRIPTION:
The objective of the present study was to determine the effects of high-intensity interval training on cognitive flexibility among female teenagers. The current study suggests that the high intensity physical training improves the cognitive ability of the participants. Evidence indicates that regular physical activity and high intensity interval training improves the physical strengthening and corresponding improvements in cardiopulmonary physical fitness that results in the increase in cerebral perfusion and vasoreactivity across the human lifespan. The betterment in the cerebral perfusion leads to better cognitive ability and mental health.

The physical activity program comprises 8 weeks consisting of Low-intensity interval training in the first week to high-intensity interval training in the 8th week. Participants of the two groups i.e., experimental and control groups were assessed at baseline fourth and eighth week by Digital Span and Mini mental state examination.

The current study from the statistical analysis suggests that better results are obtained by high intensity physical activity among the female teenagers overtime both in terms of cognitive ability and physical strength.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * Female gender only
  * Age 13-19 years of female teenagers
  * Absence of serious medical or mental illness
  * volunteered to participate in this study

Exclusion Criteria:

* Participants failing to fall in this category would be excluded from the study. Diagnosed Psychiatric illness Acute or Chronic Pain and Infections Known case of bone fragility Unstable cardiovascular disease Severe cognitive, visual, or auditory impairment

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female Teenagers
Enrollment: 40 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Digit Span (DGS) | Baseline to 8 weeks
  Cognitive Flexibilty was assessed by Digit Span (DGS), is a measure of verbal short-term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span. This is a verbal task, with stimuli presented auditory, and responses spoken by the participant and scored accordingly
Mini Mental State Examination (MMSE) | Baseline to 8 weeks
  The MMSE is a brief screening tool that provides a quantitative assessment of cognitive impairment and records cognitive changes over time (23). The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Faculty of Rehabilitation & Allied Health Sciences, Riphah International University
Locations (1):
- RIPRS, Sukkur, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No